CLINICAL TRIAL: NCT07386483
Title: Strategic Timing of Resistance Training to Guard Against Antipsychotic-Induced Metabolic Syndrome (START GAAIMS): A Feasibility Study for a Prospective, Two-Arm, Randomised Controlled Trial to Evaluate the Effects of a Resistance Training Intervention on Body Composition and Metabolic Health in People With First-Episode Psychosis
Brief Title: Strategic Timing of Resistance Training to Guard Against Antipsychotic-Induced Metabolic Syndrome
Acronym: START GAAIMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: START GAAIMS; ICAT-2022-001 (Other Grant/Funding Number: Irish Clinical Academic Training Programme)
Record Dates: First submitted 2026-01-09; First posted 2026-02-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training programme + Treatment as usual (Experimental): Participants will receive a 12-week, twice-weekly supervised resistance training programme, as well as their usual care from their community early intervention in psychosis team.
  Interventions: Other: Resistance training programme
- Treatment as Usual (No Intervention): This arm will receive the standard care from their community early intervention in psychosis team. After 12 weeks, they will be offered the 12-week, twice weekly resistance training programme

INTERVENTIONS:
Other: Resistance training programme — Participants will attend a 12-week supervised resistance training programme consisting of two 60-minute sessions per week. Each session includes a 5-10 minute aerobic warm-up, 45-50 minutes of resistance exercises, and a 5-minute cool-down. The programme is individualised and supervised by a qualified exercise practitioner.
  The intervention targets major muscle groups using 6-8 core exercises (e.g., chest press, lat pulldown, leg press, seated row, overhead press) performed in 3 sets of 6-12 repetitions. Training begins with resistance bands to establish technique (weeks 1-2) before progressing to machine and free weights. The principle of progressive overload is applied by increasing the weight once a participant can comfortably complete 3 sets of 10 repetitions in two consecutive sessions. Sessions are conducted in small groups to foster social support
  Arms: Resistance training programme + Treatment as usual

SUMMARY:
This study is evaluating whether a supervised resistance training (strength training) programme is feasible to perform in a first-episode psychosis service. It is also evaluating if resistance training can prevent harmful weight gain and improve physical health in people who have recently been diagnosed with First-Episode Psychosis and are starting antipsychotic medication.

Antipsychotic medications are essential for treating psychosis, but they frequently cause rapid weight gain and metabolic side effects (such as changes in blood sugar and cholesterol) within the first few months of treatment. Resistance training is a form of exercise that builds muscle and improves how the body uses energy. An excess of calories, which would otherwise lead to accumulation of fat (adipose tissue), can help build strength and increase muscle size when paired with resistance training.

Participants in this study will be randomly assigned to one of two groups:

Intervention Group: Participants will receive their standard medical care plus a 12-week resistance training programme. This involves attending two 60-minute exercise sessions per week, supervised by a qualified instructor. The sessions will include exercises using resistance bands, machine weights, and free weights tailored to the individual's ability.

Control Group: Participants will receive standard medical care only for the first 12 weeks.

The study uses a "crossover" design, which means that after the initial 12 weeks, the Control Group will be offered the same 12-week resistance training programme.

The main goals of this study are to determine if it is feasible to run this type of exercise programme for this group of patients and to measure the effects of the training on body fat levels, muscle strength, and overall physical and mental health

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, a participant must meet the following criteria:

1. Aged between 18 and 65 years.
2. Has the capacity to provide written informed consent.
3. Has a clinical diagnosis of a First-Episode Psychosis (affective or non-affective) made within the past three months.
4. Has had a cumulative lifetime exposure to antipsychotic medication for less than four weeks at the time of enrolment.
5. Be prescribed an antipsychotic medication at the time of enrolment.
6. Every effort will be made to include the migrant population, who have double the risk of developing psychosis compared to the general population. An interpreter service will be used during the consent stage to ensure fully informed consent is established.

Exclusion Criteria

A participant will be excluded from the study if they meet any of the following criteria:

1a. A medical condition that, in the investigator's opinion, would prevent them from giving informed consent.

1b. A medical condition that, in the investigator's opinion, would prevent them from safely participating in an exercise programme (e.g., severe, unstable cardiovascular disease, significant musculoskeletal injury).

2. Pregnant women will not be included, as hormonal changes would increase the risk of musculoskeletal injury (due to relaxin increasing laxity in ligaments and joints), maternal and foetal cardiovascular strain during the Valsalva manouevre, and additional confounders (due to pregnancy's effects on metabolism, energy levels, and physical capacity). Pregnancy is also associated with changes in body composition which affect the measurement of the primary outcome.

3. Currently participating in another clinical trial of an investigational medicinal product or device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in body fat percentage | Baseline, 12 weeks
  Body composition will be assessed using a Tanita mc-780MA body composition analyser. The outcome measure is the difference in the change in body fat percentage between the intervention and control groups
Number of participants recruited | Baseline, 12 weeks, 24 weeks
  Feasibility will be determined by achieving the target of 40 participants over the 24-month recruitment period.
Attendance by participants to intervention | Baseline, 12 weeks, 24 weeks
  Feasibility will be measured by adherence to the intervention: Determined by the percentage of participants randomised to the intervention arm who complete at least 16 of the 24 supervised sessions (≥66% adherence). The intervention is considered deliverable if ≥66% of participants meet this threshold.

SECONDARY OUTCOMES:
Body Mass Index | Baseline, 12 weeks, 24 weeks
  Assessment of Body Mass Index (BMI, kg/m²) will be calculated by combining weight, measured with Tanita mc-780MA body composition analyser, and height, measured with a wall mounted height measurer.
Weight | Baseline, 12 weeks, 24 weeks
  Measured with Tanita mc-780MA body composition analyser. Will be used in conjunction with height to estimate Body Mass Index
Change in HDL | Baseline, 12 weeks, 24 weeks
  Assessment of fasting blood samples to evaluate High-Density Lipoprotein (HDL) cholesterol
Change in Muscular Strength (Upper and Lower Body) | Baseline, 12 weeks, 24 weeks
  Maximal strength will be assessed using the One Repetition Maximum or Three Repitition Maximum test for the Chest Press, Row, and Leg Press exercises.
Change in LDL | Baseline, 12 weeks, 24 weeks
  Assessment of fasting blood samples to evaluate Low-Density Lipoprotein (LDL) cholesterol
Changes in fasting glucose | Baseline, 12 weeks, 24 weeks
  Assessment of fasting blood samples to evaluate Glucose
Change in HbA1c | Baseline, 12 weeks, 24 weeks
  Assessment of blood samples to evaluate Glycated Haemoglobin (HbA1c), which measures average blood glucose levels over the past 2-3 months by checking sugar attached to red blood cells. It is used to diagnose prediabetes (42-47) mmol/mol and diabetes (48) mmol/mol.
Change in functioning | Baseline, 12 weeks, 24 weeks
  Change in clinician-rated Global Assessment of Functioning (GAF) scale. On a scale of 1-100, where 100 represents superior functioning with no symptoms, and 1 represents persistent danger of severely hurting self/others or, inability to maintain minimal personal hygiene.
Change in self-rated function | Baseline, 12 weeks, 24 weeks
  Change in scores of the patient-rated 5-level EQ-5D version (EQ-5D-5L). This assesses five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) across five levels of severity, providing a sensitive, validated tool for clinical and economic research.
  Consists of the EQ-5D descriptive system (5-digit health state) and the EQ VAS (Visual Analogue Scale), which records self-rated health on a 0-100 scale.
  Scoring: Results are used to create utility values (index scores) anchored at 0 (dead) and 1 (full health)
Change in recovery scale scores | Baseline, 12 weeks, 24 weeks
  Change in score of the Questionnaire about the Process of Recovery, a 15-item self-administered tool used to measure personal recovery in individuals with mental health conditions, particularly psychosis. Items are rated on a 5-point Likert scale, ranging from 0 (strongly disagree) to 4 (strongly agree).
  Higher total scores indicate a greater degree of personal recovery
Change in psychiatric symptoms | Baseline, 12 weeks, 24 weeks
  Assessment of psychiatric symptoms using Brief Psychiatric Rating Scale (BPRS). Clinicians rate each symptom construct on a scale usually ranging from 1 (not present) to 7 (extremely severe), meaning a higher total score indicates greater psychopathology
Height | Baseline, 12 weeks, 24 weeks
  Measured with a wall mounted height measurer. Note, height is not expected to change, but will be used in order to calculate Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Brian O'Donoghue, MD, PhD, Principal Investigator — University College Dublin
Locations (1):
- St Vincent's University Hospital / University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data (IPD) will be made available to researchers upon reasonable request following the publication of the main trial results. In accordance with FAIR data principles, the study data will be stored securely, and all data analysis will be performed in R, with the analysis code also made available to ensure reproducibility.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Protocol - Immediately Analytic code and CSR - Upon completion of study - anticipated April 2028
Access Criteria: Principal Investigators of separate studies will be allowed to access the IPD upon reasonable request
URL: https://progressresearch.org/our-projects/